CLINICAL TRIAL: NCT02564276
Title: Indocyanine Green Versus Blue Dye for Detection of Sentinel Lymph Node In Endometrial Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CE 15.114
Record Dates: First submitted 2015-09-29; First posted 2015-09-30 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2016-06

CONDITIONS: Endometrial Neoplasms
Keywords: Indocyanine Green; Sentinel Lymph Node Biopsy
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Indocyanine Green on the right side (Experimental): Indocyanine Green will be injected on the right side of the cervix and Methylene blue on the left side of the cervix.
  Interventions: Procedure: Sentinel lymph node biopsy
- Methylene Blue on the right side (Experimental): Methylene blue will be injected on the right side of the cervix and Indocyanine Green on the left side of the cervix.
  Interventions: Procedure: Sentinel lymph node biopsy

INTERVENTIONS:
Procedure: Sentinel lymph node biopsy

SUMMARY:
To determine the difference in the proportion of hemipelves with successful detection of Sentinel Lymph Node according to the dye used (indocyanine green with near-infrared imaging vs blue dye) in women with endometrial cancer.

DETAILED DESCRIPTION:
In the past few years, Sentinel Lymph Node (SLN) procedure has emerged as an interesting solution to the debate on lymphadenectomy in endometrial cancer. Using blue-dye is inexpensive but results in an unsatisfactory detection rate of SLN. IndoCyanine Green (ICG) with near-infrared imaging is a novel technology for SLN mapping and initial reports on the use of ICG have shown high detection rate. In the present study, we aim to determine precisely the increase in detection rate of SLN associated with the use of ICG instead of blue dye. This randomized controlled trial will include patients with preoperative stage I endometrial carcinoma. All included women will undergo SLN mapping with blue dye in one hemipelvis and ICG in the other hemipelvis. Randomization will concern the side of the hemipelvis in which blue dye vs ICG mapping is used, so that the patient's contralateral hemipelvis will serve as a control to her ipsilateral hemipelvis. The primary endpoint is the difference in the proportion of hemipelves with successful detection of SLN according to the dye used. The unique precise information gained from the present study will contribute to determine whether the benefit of the use of ICG over blue dye is sufficient to justify the expense of its use.

ELIGIBILITY:
Inclusion Criteria:

* all patients with endometrial carcinoma proven by endometrial biopsy or curettage AND
* preoperative FIGO (International Federation of Gynecology and Obstetrics) stage I AND
* intended for staging via laparoscopic or robotic surgery AND
* Patients must be older than 18 year-old, able to read French or English.

Exclusion Criteria:

* preoperative FIGO stages II to IV
* previous pelvic or paraaortic lymphadenectomy or radiotherapy
* surgery that could change the uterine lymphatic drainage (myomectomy)
* iodine allergy
* pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2016-02; Primary Completion 2017-04 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
the difference in the proportion of hemipelves with successful detection of SLN according to the dye used | at time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Béatrice Cormier, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier Universitaire Montréal Hôpital Saint Luc, Montreal, Quebec, Canada

REFERENCES:
- [Result] Creasman WT, Morrow CP, Bundy BN, Homesley HD, Graham JE, Heller PB. Surgical pathologic spread patterns of endometrial cancer. A Gynecologic Oncology Group Study. Cancer. 1987 Oct 15;60(8 Suppl):2035-41. doi: 10.1002/1097-0142(19901015)60:8+3.0.co;2-8. PMID 3652025
- [Result] Abu-Rustum NR, Alektiar K, Iasonos A, Lev G, Sonoda Y, Aghajanian C, Chi DS, Barakat RR. The incidence of symptomatic lower-extremity lymphedema following treatment of uterine corpus malignancies: a 12-year experience at Memorial Sloan-Kettering Cancer Center. Gynecol Oncol. 2006 Nov;103(2):714-8. doi: 10.1016/j.ygyno.2006.03.055. Epub 2006 Jun 5. PMID 16740298
- [Result] Dankert J, Bouma J. Recurrent acute leg cellulitis after hysterectomy with pelvic lymphadenectomy. Br J Obstet Gynaecol. 1987 Aug;94(8):788-90. doi: 10.1111/j.1471-0528.1987.tb03728.x. PMID 3663535
- [Result] Querleu D, Leblanc E, Cartron G, Narducci F, Ferron G, Martel P. Audit of preoperative and early complications of laparoscopic lymph node dissection in 1000 gynecologic cancer patients. Am J Obstet Gynecol. 2006 Nov;195(5):1287-92. doi: 10.1016/j.ajog.2006.03.043. Epub 2006 May 3. PMID 16677594
- [Result] Barlin JN, Khoury-Collado F, Kim CH, Leitao MM Jr, Chi DS, Sonoda Y, Alektiar K, DeLair DF, Barakat RR, Abu-Rustum NR. The importance of applying a sentinel lymph node mapping algorithm in endometrial cancer staging: beyond removal of blue nodes. Gynecol Oncol. 2012 Jun;125(3):531-5. doi: 10.1016/j.ygyno.2012.02.021. Epub 2012 Feb 22. PMID 22366409
- [Result] Desai PH, Hughes P, Tobias DH, Tchabo N, Heller PB, Dise C, Slomovitz BM. Accuracy of robotic sentinel lymph node detection (RSLND) for patients with endometrial cancer (EC). Gynecol Oncol. 2014 Nov;135(2):196-200. doi: 10.1016/j.ygyno.2014.08.032. Epub 2014 Aug 28. PMID 25175452
- [Result] Cormier B, Rozenholc AT, Gotlieb W, Plante M, Giede C; Communities of Practice (CoP) Group of Society of Gynecologic Oncology of Canada (GOC). Sentinel lymph node procedure in endometrial cancer: A systematic review and proposal for standardization of future research. Gynecol Oncol. 2015 Aug;138(2):478-85. doi: 10.1016/j.ygyno.2015.05.039. Epub 2015 Jun 3. PMID 26047592
- [Result] Ballester M, Dubernard G, Lecuru F, Heitz D, Mathevet P, Marret H, Querleu D, Golfier F, Leblanc E, Rouzier R, Darai E. Detection rate and diagnostic accuracy of sentinel-node biopsy in early stage endometrial cancer: a prospective multicentre study (SENTI-ENDO). Lancet Oncol. 2011 May;12(5):469-76. doi: 10.1016/S1470-2045(11)70070-5. Epub 2011 Apr 12. PMID 21489874